CLINICAL TRIAL: NCT04764162
Title: Short Term Choline Supplementation and Cardiometabolic Health in Adults
Brief Title: Choline and Cardiometabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kevin Davy, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 25-521; R21AG067380 (NIH)
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Risk Factor
Keywords: insulin sensitivity; vascular function; blood pressure; continuous glucose monitoring; trimethylamine N-oxide (TMAO)
MeSH Terms: conditions — Insulin Resistance | interventions — Choline

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, crossover design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choline, then Placebo (Experimental): Participants will consume 1000 mg (2 x 500 mg) of choline supplement per day for 4 weeks, including post-testing sessions. A 2-week washout period will follow the first intervention. Then the participants will consume 1000 mg (2 x 500 mg) of placebo per day for 4 weeks, including post-testing sessions.
  Interventions: Dietary Supplement: Choline; Dietary Supplement: Placebo
- Placebo, then Choline (Experimental): Participants will consume 1000 mg (2 x 500 mg) of placebo per day for 4 weeks, including post-testing sessions. A 2-week washout period will follow the first intervention. Then the participants will consume 1000 mg (2 x 500 mg) of choline supplement per day for 4 weeks, including post-testing sessions.
  Interventions: Dietary Supplement: Choline; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Choline — 1000 mg (2 x 500 mg) choline bitartrate capsules (over-the-counter supplement)
Dietary Supplement: Placebo — Choline-matched 1000 mg (2 x 500 mg) placebo (maltodextrin) capsules

SUMMARY:
Trimethylamine-N-oxide (TMAO), a metabolite produced by gut microbial metabolism of dietary choline, has recently been causally linked to atherosclerosis in animal models and has been shown to be predictive of cardiovascular disease (CVD) risk in some but not all cohort studies. The relevance of observations in animals to humans is unclear and little information is available on the mechanisms linking TMAO to increased CVD risk. Vascular dysfunction plays a critical role in the initiation and progression of atherothrombotic disease. Whether TMAO impairs vascular function in humans is not known. The purpose of this study is to determine if short term supplementation of dietary choline, which increases TMAO, affects CVD risk factors, such as glucose homeostasis and vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-79 years
* Weight stable for previous 6 months (+2.0kg)
* Sedentary to recreationally active (<30 min aerobic exercise <2x/wk)
* No plans to gain/lose weight or change physical activity level
* Verbal and written informed consent
* Willing to be randomized to treatment order
* Fully vaccinated against COVID-19

Exclusion Criteria:

* BMI > 35 kg/m2
* Smoking
* Pregnant or plans of becoming pregnant
* Vegetarian or Vegan
* Changed dietary patterns within the last month
* Diabetes (or use of diabetes medications) or unstable heart disease
* Untreated high blood pressure or high cholesterol
* Health problems that mide it unsafe to participate
* Taking medications, vitamins or supplements that could affect study outcomes (including but not limited to aspirin, antibiotics, prebiotics, and probiotics)
* Known allergy, hypersensitivity, intolerance to choline supplement or its ingredients
* Trimethylaminuria or "fish odor" syndrome

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Davy, PhD, Principal Investigator — Virginia Polytechnic Institute & State University
Locations (1):
- Virginia Polytechnic and State University, Blacksburg, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 individuals were screened and 10 were randomized. Those not randomized voluntarily withdrew from the study.
Pre-assignment Details: 4 enrolled participants voluntarily withdrew from the study and did not complete any pre-testing sessions before their first assigned intervention.
Period: Overall Study
Arm/Group | Choline, Then Placebo | Placebo, Then Choline
Started | 3 | 7
Completed | 3 | 6
Not Completed | 0 | 1
Not completed — Did not complete oral glucose tolerance tests due to low BP. Did complete other study measures. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Choline, Then Placebo | Placebo, Then Choline | Total
Number analyzed (Participants) | 3 | 7 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (16) | 50 (17) | 48 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 7 | 10
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 28.3 (3.4) | 24.2 (2.96) | 25.5 (3.5)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 121 (9) | 119 (14) | 120 (13)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 75 (9) | 72 (6) | 73 (7)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 113 (63) | 117 (66) | 116 (62)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 183 (36) | 200 (35) | 195 (34)
HDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 42 (3) | 55 (20) | 51 (17)
LDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 120 (22) | 122 (22) | 121 (21)
Glucose [Mean (Standard Deviation); unit: mg/dL] | 95 (2) | 90 (5) | 92 (5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Insulin Sensitivity at 4 Weeks
Description: Participants will complete a 2-hour glucose tolerance test at baseline, immediately following the first intervention, after a 2-week washout, and immediately following the second intervention. A catheter will be placed in one of the participant's arms. After a baseline blood draw to measure fasting levels of glucose, insulin, cholesterol and other factors, participants will drink a glucose beverage (75 g). Blood will be collected in small amounts (less than one half teaspoon) at eight timepoints over a 2-hour period. Insulin sensitivity will be calculated using Matsuda's index (a ratio with no units). This test will be conducted two times separated by about 4 weeks for each intervention (choline, placebo).
Time Frame: Calculated difference between the baseline and 4-week testing session for each intervention
Population: All participants received each supplementation intervention during their respective cross-over randomization assignment. Therefore, Outcome Measures are reported per intervention.
Measure: Mean (Standard Deviation); unit: Calculated Ratio - No units
Groups:
- Choline: Participants will consume 1000 mg (2 x 500 mg) of choline per day for 4 weeks, including post-testing sessions.
- Placebo: Participants will consume 1000 mg (2 x 500 mg) of placebo (maltodextrin) per day for 4 weeks, including post-testing sessions.
Arm/Group | Choline | Placebo
Number analyzed (Participants) | 9 | 9
Calculated Ratio - No units | 0.28 (0.8) | -0.29 (0.45)

2. Secondary Outcome: Change in 24-hour Area Under the Curve for Glucose Levels After Supplementation
Description: Glucose will be monitored by a Continuous Glucose Monitor (CGM) sensor (Enlite Sensor; Medtronic, Inc. or FreeStyle Libre Pro; Abbott) and this will be placed on the participant's abdomen or back of the upper arm in order to measure glucose continuously. The measured glucose levels will be assessed by an iPro2 Professional CGM; Medtronic, Inc. or FreeStyle Libre Pro reader; Abbott; and the CGM will be worn for 4 consecutive days. This test will be conducted two times separated by about 4 weeks for each intervention (choline, placebo).
Time Frame: Difference in 24-hour glucose levels during free living at baseline and 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL per day
Arm/Group | Choline | Placebo
Number analyzed (Participants) | 9 | 9
mg/dL per day | 7032.5 (10709.5) | -2685 (17213.2)

ADVERSE EVENTS:
Time Frame: 10 weeks total: 4 weeks for each intervention, 2-week washout between interventions
Description: All participants who received at least one dose of intervention were supervised for safety.
Groups:
- Choline: Participants will consume 1000 mg (2 x 500 mg) of choline supplement per day for 4 weeks, including post-testing sessions.
- Placebo: Participants will consume 1000 mg (2 x 500 mg) of placebo per day for 4 weeks, including post-testing sessions.
Arm/Group | Choline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT04764162/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT04764162/ICF_000.pdf